CLINICAL TRIAL: NCT03524937
Title: Prevention of Delirium in Intensive Care by Melatonin: a Prospective, Multicentre, Randomized, Double Blind, Placebo, Multi-arm, Multi-stage Study
Brief Title: Prevention of Delirium in Intensive Care by Melatonin
Acronym: DEMEL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P160942J
Record Dates: First submitted 2018-04-25; First posted 2018-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Mechanically Ventilated Patients
Keywords: Delirium; Mechanical ventilation; Intensive care unit; Prevention; Pharmacokinetics; Melatonin
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MELATONIN (LOW DOSE) (Experimental): Daily administration of melatonin by enteral route at 0.3 mg/day (low dose arm), up to 14 days.
  Interventions: Drug: MELATONIN (LOW DOSE)
- MELATONIN (HIGH DOSE) (Experimental): Daily administration of melatonin by enteral route at 3 mg/day (high dose arm), up to 14 days.
  Interventions: Drug: MELATONIN (HIGH DOSE)
- PLACEBO (Placebo Comparator): Daily administration of identical placebo up to 14 days.
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: MELATONIN (HIGH DOSE) — Enteral melatonin (3mg) will be given at 21:00h daily, starting on the day of enrolment until ICU discharge, death, or up to 14 days
  Other Names: N-acetyl-5-methoxytryptamine
  Arms: MELATONIN (HIGH DOSE)
Drug: MELATONIN (LOW DOSE) — Enteral melatonin (0.3mg ) will be given at 21:00h daily, starting on the day of enrolment until ICU discharge, death, or up to 14 days
  Other Names: N-acetyl-5-methoxytryptamine
  Arms: MELATONIN (LOW DOSE)
Drug: PLACEBO — Study drug will be given at 21:00h daily, starting on the day of enrolment until ICU discharge, death, or up to 14 days.
  Arms: PLACEBO

SUMMARY:
This is a double-blind, randomized, placebo-controlled, Phase 2b/3 two-part adaptive clinical trial. The trial is designed to investigate the pharmacokinetics and the efficacy of multiple dosing regimens of melatonin and to confirm the efficacy and safety of one dosing regimen in prevention for delirium.

DETAILED DESCRIPTION:
Treatment of the study is a single daily fixed-hour (21h) dose of 15 mL of an oral syrup, at one of the 3 following concentrations of melatonin: 0 mg/ml i.e. 0 mg/day (placebo); 0.02 mg/ml, i.e. 0.3 mg/day (low dose of melatonin) or 0.2 mg/ml, i.e. 3 mg/day (high dose of melatonin). The three dosages will be identical in appearance and volume.Treatment will be administered up to Day-14 (or death or discharge if these occur before Day-14). Randomization will be stratified by center.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient under invasive mechanical ventilation
* Anticipated stay in intensive care unit of at least 48 hours
* Informed consent signed by the patient or a relative or emergency consent

Exclusion Criteria:

* Invasive mechanical ventilation for more than 48 hours
* known pregnancy or breastfeeding
* No understanding of the French language, deafness
* Dementia (Mini Mental State <20) or known chronic psychosis
* Delirium (positive CAM-ICU score) before or at the time of randomization
* Alcohol withdrawal syndrome before or at the time of randomization with Cushman score ≥5
* Inability to use the enteral route, food intolerance with vomiting
* Severe hepatic insufficiency (prothrombin level <30%)
* Ongoing treatment with melatonin or a drug that interacts or modifies its metabolism (fluvoxamine, 5- or 8-methoxypsoralen, estrogen, cimetidine, carbamazepine, rifampicin)
* known allergy to melatonin
* moribund state
* Patient admitted to intensive care for cardiopulmonary arrest, stroke, head trauma, neurosurgery.
* Patient not affiliated to social security
* Patient participating in another interventional clinical study with melatonin and / or for whom delirium is the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Delirium incidence | up to 14 days

SECONDARY OUTCOMES:
Day 28 Mortality | at day 28
  Day 28 Mortality
Hospital mortality | At day 28
  Hospital mortality
ICU mortality | at day 28
  ICU mortality
Evaluate number of days alive without coma nor delirium | Up to day 14
  days alive without coma nor delirium
Duration of delirium | 14 days
  Duration of delirium
Duration of mechanical ventilation | Up to day 28
  Duration of mechanical ventilation
Hospital length of stay | at day 28
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: France GUYOT, Study Chair — DRCI-Assistance Publique des Hopitaux de paris
Locations (1):
- Henri-Mondor Hospital, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Derived] Mekontso Dessap A, Ricard JD, Contou D, Desnos C, Decavele M, Sonneville R, Vivier E, Terzi N, Callahan JC, Jochmans S, Leon R, Carreira S, Nseir S, Chemouni F, Castelain V, Paul M, Benoist JF, Audureau E, Razazi K; CARMAS and the REVA research networks, on behalf of the DEMEL Investigators. Melatonin for prevention of delirium in patients receiving mechanical ventilation in the intensive care unit: a multiarm multistage adaptive randomized controlled clinical trial (DEMEL). Intensive Care Med. 2025 Jul;51(7):1292-1305. doi: 10.1007/s00134-025-08002-z. Epub 2025 Jul 3. PMID 40608082